CLINICAL TRIAL: NCT00937456
Title: Open vs Laparoscopically-assisted Esophagectomy for Cancer: A Multicentric Phase III Prospective Randomized Controlled Trial
Brief Title: Open Versus Laparoscopically-assisted Esophagectomy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008_24/0904; PHRC 2008/1907 (Other: DHOS); 2009-A00144-53. (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Esophageal Cancer
Keywords: Esophagus; Cancer; Surgery; Laparoscopy; Randomized trial; Esophageal cancer deemed to be resectable
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopically-assisted esophagectomy (Experimental): Laparoscopically-assisted esophagectomy: standard abdominal procedure of gastric mobilisation but through laparoscopic route. Right thoracotomy as usual.
  Interventions: Procedure: Laparoscopically-assisted esophagectomy
- Open esophagectomy (Active Comparator): Conventional open esophagectomy: Esophagectomy with extended 2-field lymphadenectomy through laparotomy and right thoracotomy (Ivor-Lewis standard procedure)
  Interventions: Procedure: Laparoscopically-assisted esophagectomy

INTERVENTIONS:
Procedure: Laparoscopically-assisted esophagectomy — To compare during the abdominal approach the laparoscopic route to the open route for gastric mobilization. Thoracic approach will be the same between the 2 arms through thoracotomy with extended two field lymphadenectomy
  Other Names: esophagectomy with extended two-field lymphadenectomy

SUMMARY:
To compare laparoscopically-assisted gastric mobilization versus open gastric mobilization in Ivor-Lewis esophagectomy for esophageal cancer, with open thoracic approach in the 2 arms.

DETAILED DESCRIPTION:
Open Versus Laparoscopically-assisted Esophagectomy for Cancer

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell or adenocarcinoma of the thoracic esophagus T1, T2, T3, N0-N1, M0, before any treatment
* Middle or lower third esophageal carcinoma, junctional tumor Siewert type I
* Patients who underwent or not neoadjuvant chemotherapy or chemoradiation
* Tumor deemed to be resectable in a curative intent at the preoperative setting
* Age less than 75 years old, OMS status 0, 1 or 2
* Patient who can undergo one or the other surgical modality
* Written informed consent form
* Possible follow-up

Exclusion Criteria:

1. General criteria: PO2 ≤ 60 mmHg; PCO2 > 45 mmHg; FEV ≤ 1000 ml/sec

   * Hepatic cirrhosis
   * Recent myocardial infarction (in the previous 6 months) or progressive coronary disease
   * Distal arteritis (Leriche-Fontaine stage II upwards)
   * Concomitant cancer, other than subcarinal esophageal cancer
2. Disease-related factors

   * Invasion of subclavicular lymph nodes in a clinical examination or on biospy
   * Lymph nodes near the origin of the celiac artery with a diameter ≥ 1 cm on CT or that appear to be suspect on endoscopic ultrasound (to differentiate them from the paracardial or left gastric lymph nodes, which does not constitute an exclusion criterion)
   * Recurrent nerve palsy
   * Evidence of extension to the tracheobronchial tree
   * Signs of mediastinal invasion (vertebral contact, aortic contact ≥ 90°, or invasion of nonresectable neighboring organs such as the aorta, trachea, main bronchi, etc.)
   * Distant metastasis
3. Laparoscopy-related factors

   * Patient presenting a general contraindication to laparoscopy
   * A history of median or subcostal laparotomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-10-07; Primary Completion 2011-10 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
To decrease postoperative major 30-days morbidity from 45% in the open arm to 25% in the laparoscopically-assisted arm. | 30 days

SECONDARY OUTCOMES:
overall morbidity | 30 days
disease free survival | 2 years
overall survival | 2 years
quality of life | 2 years
economical interest of the surgical technique apprehended through a hospital point of view | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariette, MD, PhD, Principal Investigator — University Hospital of Lille, France
Locations (11):
- France (11):
  - Hopital Du Haut Leveque, Bordeaux
  - Hopital Ambroise Pare Ap-Hp, Boulogne-Billancourt
  - Hotel Dieu, Clermont-Ferrand
  - Hopital Louis Mourier, Colombes
  - Hopital de La Croix Rousse, Lyon
  - Hopital St Marguerite Ap-Hm, Marseille
  - Hopital St Louis Ap-Hp, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hopitalpontchaillou, Rennes
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Hopital Purpan, Toulouse

REFERENCES:
- [Derived] Nuytens F, Dabakuyo-Yonli TS, Meunier B, Gagniere J, Collet D, D'Journo XB, Brigand C, Perniceni T, Carrere N, Mabrut JY, Msika S, Peschaud F, Prudhomme M, Markar SR, Piessen G; Federation de Recherche en Chirurgie (FRENCH) and French Eso-Gastric Tumors (FREGAT) Working Groups. Five-Year Survival Outcomes of Hybrid Minimally Invasive Esophagectomy in Esophageal Cancer: Results of the MIRO Randomized Clinical Trial. JAMA Surg. 2021 Apr 1;156(4):323-332. doi: 10.1001/jamasurg.2020.7081. PMID 33595631
- [Derived] Mariette C, Markar SR, Dabakuyo-Yonli TS, Meunier B, Pezet D, Collet D, D'Journo XB, Brigand C, Perniceni T, Carrere N, Mabrut JY, Msika S, Peschaud F, Prudhomme M, Bonnetain F, Piessen G; Federation de Recherche en Chirurgie (FRENCH) and French Eso-Gastric Tumors (FREGAT) Working Group. Hybrid Minimally Invasive Esophagectomy for Esophageal Cancer. N Engl J Med. 2019 Jan 10;380(2):152-162. doi: 10.1056/NEJMoa1805101. PMID 30625052
- [Derived] Briez N, Piessen G, Bonnetain F, Brigand C, Carrere N, Collet D, Doddoli C, Flamein R, Mabrut JY, Meunier B, Msika S, Perniceni T, Peschaud F, Prudhomme M, Triboulet JP, Mariette C. Open versus laparoscopically-assisted oesophagectomy for cancer: a multicentre randomised controlled phase III trial - the MIRO trial. BMC Cancer. 2011 Jul 23;11:310. doi: 10.1186/1471-2407-11-310. PMID 21781337